CLINICAL TRIAL: NCT02297178
Title: A Follow-net Investigation of a Randomised Study of Cystoscopy and Urethral Dilatation Versus Cystoscopy Alone in Women With Overactive Bladder Syndrome and Impaired Voiding
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit resaerch staff for study
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Jonathan Duckett, Consultant Gynaecologist and Obstetrician, Medway NHS Foundation Trust
Other Study IDs: MedwayUD
Record Dates: First submitted 2014-11-11; First posted 2014-11-21 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Overactive Bladder; Voiding Dysfunction; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Cystoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystoscopy Alone: Patients who received cystoscopy only for treatment of OAB and voiding dysfunction.
  Interventions: Procedure: Cystoscopy only
- Cystoscopy & Urethral Dilatation: Patients who received urethral dilatation and cystoscopy for treatment of OAB and voiding dysfunction.
  Interventions: Procedure: Cystoscopy and Urethral dilatation

INTERVENTIONS:
Procedure: Cystoscopy only — Cystoscopy performed for investigation and treatment of OAB and voiding dysfunction
  Groups: Cystoscopy Alone
Procedure: Cystoscopy and Urethral dilatation — Cystoscopy and urethral dilatation performed for investigation and treatment of OAB and voiding dysfunction
  Groups: Cystoscopy & Urethral Dilatation

SUMMARY:
Urinary incontinences is a highly prevalent and distressing condition which has a significant impact on health related quality of life in millions of women worldwide. Of all women with incontinence, 90% will have overactive bladder symptoms (OAB), and 50% will have detrusor overactivity (DO) on cystometry. The overactive bladder syndrome is defined by the International Continence society as "Urinary urgency, with or without urge incontinence, usually with frequency and nocturia if there is a no infection or proven pathology" (Abrams et al 2002)

Initial management of OAB and DO consists of conservative measures such as altering fluid intake, bladder retraining and drug therapy. The next step consists of interventions such as cystoscopy and urethral dilatation, on the basis that it will allow intrinsic bladder problems such as interstitial cystitis to excluded, excluded, and may confer a symptomatic benefit.

The original study showed no benefit of urethral dilatation versus no dilatation at 6 months follow up (Duckett 2007). The investigators do not know the natural history of patients with voiding dysfunction. Therefore reviewing their symptoms will give a better idea of what happens to these patients symptoms over time.

DETAILED DESCRIPTION:
Urinary incontinences is a highly prevalent and distressing condition which has a significant impact on health related quality of life in millions of women worldwide. Of all women with incontinence, 90% will have overactive bladder symptoms (OAB), and 50% will have detrusor overactivity (DO) on cystometry. The overactive bladder syndrome is defined by the International Continence society as "Urinary urgency, with or without urge incontinence, usually with frequency and nocturia if there is a no infection or proven pathology" (Abrams et al 2002)

Initial management of OAB and DO consists of conservative measures such as altering fluid intake, bladder retraining and drug therapy. The next step consists of interventions such as cystoscopy and urethral dilatation, on the basis that it will allow intrinsic bladder problems such as interstitial cystitis to excluded, excluded, and may confer a symptomatic benefit.

Cystoscopy and urethral dilatation have long been advocated as empirical treatments for women with lower urinary tract symptoms (LUTS). A review of the literature reveals a marked lack of evidence regarding the survey of practice amongst UK urologists found that 61% had performed urethral dilatation 7 or more times during the year in which the survey was conducted, although 55% believed that less than half of the patients experience long term improvement (Masarani and Willis, 2006)

The original study showed no benefit of urethral dilatation versus no dilatation at 6 months follow up (Duckett 2007). The investigators do not know the natural history of patients with voiding dysfunction. Therefore reviewing their symptoms will give a better idea of what happens to these patients symptoms over time. The aim of the study is to identify any long term benefit from urethral dilatation over cystoscopy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Significant Overactive Bladder Symptoms

   * Based on scoring 1 or 2 on the Urgency Perception Scale
   * On the symptoms domain of the KHQ
   * More than 8 voids per day on frequency volume chart +/- 2 or more episodes of nocturia
2. Pressure flow studies demonstrate a maximum flow rate of less than 15ml on a minimum voided volume of 200ml with a high or normal detrusor pressure at maximum flow or post-void residual of 200ml or over
3. Patients must be able to give informed consent for the study.

Exclusion Criteria:

1. Presence of concurrent urodynamic stress incontinence.
2. Patients with bladder pathology or haematuria of unknown origin.
3. Patients with neurological disorders (as these may affect voiding).
4. Symptomatic pelvic organ prolapse requiring intervention
5. Patients with bladder pathology (including urinary tract infection) or haematuria of unknown origin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Entry to the study will be offered to all women previously recruited into the original randomised controlled trial. This study is a 3 year follow up of a randomised controlled trial. Patients will be sent a letter offering a review appointment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ICIQ-Fluts questionnaire | 3 years
  To identify if there is any long term benefit from urethral dilatation over cystoscopy alone. Their baseline symptoms will be assessed and compared to those identified at baseline in the previous study.

SECONDARY OUTCOMES:
King's Health Questionnaire | 3 years
  To identify if there is any long term benefit from urethral dilatation over cystoscopy alone. Their baseline symptoms will be assessed and compared to those identified at baseline in the previous study.
Urgency Perception Scale Questionnaire | 3 years
  To identify if there is any long term benefit from urethral dilatation over cystoscopy alone. Their baseline symptoms will be assessed and compared to those identified at baseline in the previous study.
Uroflowmetry | 3 years
  Flow rates will be repeated in all patients allowing for an objective comparison post-operatively and 3 years later.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan RA Duckett, FRCOG, MBChB, Principal Investigator — Medway Maritime Hospital

REFERENCES:
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Result] Duckett JR, Basu M. The predictive value of preoperative pressure-flow studies in the resolution of detrusor overactivity and overactive bladder after tension-free vaginal tape insertion. BJU Int. 2007 Jun;99(6):1439-42. doi: 10.1111/j.1464-410X.2007.06842.x. Epub 2007 Apr 5. PMID 17419703
- [Result] Masarani M, Willis RG. Urethral dilatation in women: urologists' practice patterns in the UK. Ann R Coll Surg Engl. 2006 Sep;88(5):496-8. doi: 10.1308/003588406X114884. PMID 17002859